CLINICAL TRIAL: NCT06293066
Title: Performance of Ultrasound in Women With Postmenopausal or Abnormal Uterine Bleeding Between White and Black Ethnic Groups
Brief Title: Performance of Ultrasound in Women With Postmenopausal or Abnormal Uterine Bleeding Between White and Black Ethnic Groups- a Retrospective Cohort Study.
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH23-257
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Postmenopausal Bleeding; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Usefulness of transvaginal ultrasound

SUMMARY:
Primary Objective:

To assess whether there is a higher incidence of uninformative ultrasound in black vs white women

DETAILED DESCRIPTION:
Retrospective cohort study

Study Subjects:

Women 45 years or over seen in the 'two-week wait' rapid access Gynaecology clinic with suspected endometrial cancer due to abnormal vaginal bleeding over the course of 2022. Only people with documented ethnicity will be included.

Study Procedures:

Cases will be identified by searching our two-week referral and ultrasound records . Clinical data collected includes age, BMI, previous abdominal uterine surgery (Caesarean section or open myomectomy) and parity. Symptoms will be categorised into postmenopausal bleeding with no hormone use, unscheduled bleeding on hormone replacement therapy (HRT) or abnormal perimenopausal bleeding (in women over 45 years of age).

Ultrasound data recorded will be the presence or absence of fibroids, whether transabdominal ultrasound was needed in addition to transvaginal or transrectal ultrasound, whether the endometrium could be seen clearly (i.e whether the ultrasound examination was informative) and the endometrial thickness in those where it was. Clinical outcomes recorded will be the need for endometrial sampling, mode of sampling and histology results. The local cancer registry will be checked for the year following the study to check for any subsequent cancers in women discharged without endometrial sampling.

ELIGIBILITY:
Inclusion Criteria:

* Women seen in the 'two-week wait' rapid access Gynaecology clinic with suspected endometrial cancer due to abnormal vaginal bleeding over the course of 2022

  * 45 years of age or older
  * Ethnicity documented in their clinical notes

Exclusion Criteria:

* Ethnicity data not available

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with postmenopausal bleeding referred to the gynaecology rapid access clinic
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
To assess whether there is a higher incidence of uninformative ultrasound in black vs white women | Review of patients who attended clinic in 2022
  The need for further investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Suite 8, King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided